CLINICAL TRIAL: NCT02110342
Title: A Phase One Open-Label Single-Radiolabeled Dose Study To Investigate The Absorption, Metabolism, And Excretion Of [14C] PF-04449913 In Healthy Male Volunteers
Brief Title: A Study To Understand How Radiolabelled PF-04449913 Is Taken Up By The Body, Broken Down And Then Removed From The Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B1371009
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: PF-04449913; [14C]PF-04449913; Human ADME; Radiolabel; Mass Balance; Pharmacokinetics
MeSH Terms: interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: [14C] PF-04449913

INTERVENTIONS:
Drug: [14C] PF-04449913 — Single oral dose of 100 mg PF-04449913 + 100µCi of [14C] PF-04449913

SUMMARY:
The study aims to understand, using radiolabelled PF-04449913, how this compound is modified by the body once it is absorbed. The study also aims to understand how much of the compound is broken down and how much leaves the body unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years (inclusive):Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects enrolled in a previous radionucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry.
* A positive urine drug screen or urine cotinine test
* 12 lead ECG demonstrating QTc >450 or a QRS interval >120 msec msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility. Subjects with family history of myocardial infarction, congenital long QT syndrome, torsades de pointes or clinically significant ventricular arrhythmias. Subjects should be within normal range of potassium, magnesium and calcium at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 7 days
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 7 days
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] for total radioactivity related to drug product | 7 days
  AUC (0 - 8)= Area under the plasma radioactivity concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) for total radioactivity related to drug product | 7 days
Cumulative recovery of radioactivity in excreta | 7 days
  Total percentage of dosed radioactivity recovered in urine and feces
Radioactivity in blood | 7 days
  Total percentage of radioactivity in blood related to drug product
Urine PF-04449913 PK parameters | 7 days
  Measure of renal clearance (CLr), amount excreted unchanged in urine (Ae) and the fraction of dose excreted unchanged in urine (AE%)

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 7 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Plasma Decay Half-Life (t1/2) | 7 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 7 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 7 days
  plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Madison, Wisconsin, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371009&StudyName=A%20Study%20To%20Understand%20How%20Radiolabelled%20PF-04449913%20Is%20Taken%20Up%20By%20The%20Body%2C%20Broken%20Down%20And%20Then%20Removed%20From%20The%20Body